CLINICAL TRIAL: NCT06028477
Title: Vibrotactile Coordinated Reset in Parkinson's Disease - Proof of Concept Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Vivek P. Buch, Assistant Professor of Neurosurgery, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71954
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded for 6 months followed by an unblinding of everyone with the exception of the clinical assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active stimulation (Active Comparator): Participants will receive active stimulation between 2 hours minimum and 4 hours maximum of daily vCR or sham stimulation (2 hours twice daily) at home for the first month (30 days), followed by a minimum of 1.5 hours and a maximum of 2.5 hours of daily vCR
  Interventions: Device: Stanford Glove
- Sham Stimulation (Sham Comparator): Participants will receive sham stimulation between 2 hours minimum and 4 hours maximum of daily vCR or sham stimulation (2 hours twice daily) at home for the first month (30 days), followed by a minimum of 1.5 hours and a maximum of 2.5 hours of daily vCR
  Interventions: Device: Stanford Glove

INTERVENTIONS:
Device: Stanford Glove — The non-invasive neuromodulation hardware system comprises two wireless controllers/battery packs which are fastened to the top of each hand via an adjustable elastic strap. Each controller is equipped with four vibrotactile fingertip stimulators, also known as tappers. There is a total of eight tappers (for index, middle, ring and pinkie of each hand) per system.

SUMMARY:
The purpose of our study is to evaluate Vibrotactile Coordinated Reset stimulation (vCR) and its effects on Parkinson's symptoms. vCR will be administered with a device called the Stanford Glove. vCR is expected to provide patients with a non-invasive alternative to the most widely used treatments such as Levodopa and/or deep brain stimulation. Patients will be followed for 14 months.

DETAILED DESCRIPTION:
The purpose of this study is to test the efficacy of vibrotactile coordinated reset stimulation on human subject participants with Parkinson's disease and inform the investigators on whether unilateral stimulation could be as effective as bilateral stimulation at producing clinically significant improvements in symptoms.

ELIGIBILITY:
Inclusion Criteria:

Ages 18 or older

* Diagnosed with idiopathic Parkinson's Disease
* Fluent in English
* Off-state UPDRS III motor score at least 30, as assessed within the past 6 months before study consent or at Screening Visit.
* Demonstrates understanding of the study requirements and is able and willing to sign the informed consent form and complete study procedures.

Exclusion Criteria:

* Participation in another drug, device, or biologics trial concurrently or within the preceding 30 days. Any other trial participation should be approved by the Principal Investigators.
* Pregnancy, breast-feeding or wanting to become pregnant
* Physical limitations unrelated to PD that would affect motor ratings
* Has implantation of a medical device
* Sensory abnormalities of the fingertips

Ages: 18 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in MDS-Unified Parkinson's Disease Rating Scale Part III Scale Score | Baseline and month 6
  Mean change in the MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III score.
  Minimum score - 0 indicates normal functioning Maximum score - 132 indicated severe impairment
  Lower scores indicate greater functionality and higher scores indicate severe impairment in functionality.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek P Buch, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No